CLINICAL TRIAL: NCT03880175
Title: Direct and Spillover Impacts of a Community-Level HIV/AIDS Program: Evidence From a Randomized Controlled Trial in Mozambique
Brief Title: Direct and Spillover Impacts of a Community-Level HIV/AIDS Program
Acronym: FCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Dean Yang, Professor, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00113011; AID-OAA-L-12-00001 (Other Grant/Funding Number: USAID); AID-OAA-LA-16-0004 (Other Grant/Funding Number: USAID); AID391A1500006 (Other Grant/Funding Number: USAID)
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- FCC DEB and Anti-stigma (Experimental)
  Interventions: Behavioral: FCC (Força à Comunidade e Crianças) program- direct beneficiary; Behavioral: Anti Stigma Information
- FCC DEB and HIV info (Experimental)
  Interventions: Behavioral: FCC (Força à Comunidade e Crianças) program- direct beneficiary; Behavioral: HIV/AIDS Information
- FCC DEB and ART info (Experimental)
  Interventions: Behavioral: FCC (Força à Comunidade e Crianças) program- direct beneficiary; Behavioral: ART Information
- FCC DEB and HIV-ART info (Experimental)
  Interventions: Behavioral: FCC (Força à Comunidade e Crianças) program- direct beneficiary; Behavioral: HIV/AIDS and ART Information Combined
- FCC DEB and high coupon value (Experimental)
  Interventions: Behavioral: FCC (Força à Comunidade e Crianças) program- direct beneficiary; Behavioral: High coupon value
- FCC DEB and no info (Experimental)
  Interventions: Behavioral: FCC (Força à Comunidade e Crianças) program- direct beneficiary
- FCC non-DEB and Anti-stigma (Experimental)
  Interventions: Behavioral: FCC (Força à Comunidade e Crianças) program- non-direct beneficiary; Behavioral: Anti Stigma Information
- FCC non-DEB and HIV info (Experimental)
  Interventions: Behavioral: FCC (Força à Comunidade e Crianças) program- non-direct beneficiary; Behavioral: HIV/AIDS Information
- FCC non-DEB and ART info (Experimental)
  Interventions: Behavioral: FCC (Força à Comunidade e Crianças) program- non-direct beneficiary; Behavioral: ART Information
- FCC non-DEB and HIV-ART info (Experimental)
  Interventions: Behavioral: FCC (Força à Comunidade e Crianças) program- non-direct beneficiary; Behavioral: HIV/AIDS and ART Information Combined
- FCC non-DEB and high coupon value (Experimental)
  Interventions: Behavioral: FCC (Força à Comunidade e Crianças) program- non-direct beneficiary; Behavioral: High coupon value
- FCC non-DEB and no info (Experimental)
  Interventions: Behavioral: FCC (Força à Comunidade e Crianças) program- non-direct beneficiary
- FCC control and Anti-stigma (Experimental)
  Interventions: Behavioral: Anti Stigma Information
- FCC control and HIV info (Experimental)
  Interventions: Behavioral: HIV/AIDS Information
- FCC control and ART info (Experimental)
  Interventions: Behavioral: ART Information
- FCC control and HIV-ART info (Experimental)
  Interventions: Behavioral: HIV/AIDS and ART Information Combined
- FCC control and High coupon value (Experimental)
  Interventions: Behavioral: High coupon value
- FCC control and no info (No Intervention)

INTERVENTIONS:
Behavioral: FCC (Força à Comunidade e Crianças) program- direct beneficiary — Households are directly linked to the FCC implementing organization
  Arms: FCC DEB and ART info; FCC DEB and Anti-stigma; FCC DEB and HIV info; FCC DEB and HIV-ART info; FCC DEB and high coupon value; FCC DEB and no info
Behavioral: FCC (Força à Comunidade e Crianças) program- non-direct beneficiary — Households live in FCC implementing communities but are not directly linked to the FCC implementing organization
  Arms: FCC non-DEB and ART info; FCC non-DEB and Anti-stigma; FCC non-DEB and HIV info; FCC non-DEB and HIV-ART info; FCC non-DEB and high coupon value; FCC non-DEB and no info
Behavioral: Anti Stigma Information — Adults in the households are provided anti-stigma information
  Arms: FCC DEB and Anti-stigma; FCC control and Anti-stigma; FCC non-DEB and Anti-stigma
Behavioral: HIV/AIDS Information — The households receive information about HIV infection and AIDS
  Arms: FCC DEB and HIV info; FCC control and HIV info; FCC non-DEB and HIV info
Behavioral: ART Information — The households receive information about antiretroviral therapy.
  Arms: FCC DEB and ART info; FCC control and ART info; FCC non-DEB and ART info
Behavioral: HIV/AIDS and ART Information Combined — The households receive both information about HIV/AIDS and information about antiretroviral therapy.
  Arms: FCC DEB and HIV-ART info; FCC control and HIV-ART info; FCC non-DEB and HIV-ART info
Behavioral: High coupon value — The HIV testing coupons distributed to households in this group have higher values.
  Arms: FCC DEB and high coupon value; FCC control and High coupon value; FCC non-DEB and high coupon value

SUMMARY:
The HIV/AIDS crisis in Sub-Saharan Africa has left millions of children orphaned. These children, who are potentially infected with HIV themselves, are highly vulnerable and face some serious risks to their health and overall well-being.

A variety of health and economic interventions to help orphans and vulnerable children (OVCs) (and the households in which they live) are being carried out in Mozambique by World Education Inc./Bantwana (WEI/B), funded by USAID. The program is known in Portuguese as Força à Comunidade e Crianças or FCC (in English, "Strengthening Family and Communities").

This study will collect survey and administrative data to assess the impact of the FCC program on OVCs and the households in which they live. A baseline survey was administered to define a sample of households and individuals to follow over time through the upcoming follow-up survey and to measure baseline household characteristics.

Follow-up data collection will begin in March 2019. It has several components:

1. Household survey The follow-up survey will provide measurements of the rich set of intermediate and final outcomes for the estimation of treatment effects of the FCC program.
2. Data collection on HIV testing and school attendance This study will supplement survey-reported HIV testing rates with an objective, administrative measure of HIV testing at health clinics. At the time of the follow-up survey, the survey team will recommend that eligible individuals in the household be tested for HIV at a specified local health clinic. To allow tracking of those who follow through with testing, consenting individuals will be given coupons redeemable for a small financial incentive once they have completed an HIV test.

   In addition to self-reported data on school participation by children, this study will also measure school participation directly. Both school enrollment (presence in school registration records) and school attendance (physical presence of children in school during unannounced school visits by research staff) will be measured. Project staff will visit schools in study communities to check attendance rates of specific school-aged children who were listed in the baseline survey in their community.
3. Informational treatments aimed at raising HIV testing rates To allow insight into the mechanisms through which the FCC program has its effects, this study will provide additional simple treatments in the context of the follow-up survey to explore possible FCC mechanisms: stigma reduction, HIV/AIDS information, and HIV treatment (antiretroviral therapy, or ART) information.

ELIGIBILITY:
Inclusion Criteria:

* Households that lives in one of the eligible communities.

Exclusion Criteria:

* Households that are not in the eligible communities will not be included in the survey sample.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3658 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Indicator for HIV testing coupon redemption at the household level | 14 days following the date coupons are distributed to a household.
  This is a household-level binary variable. It takes value 1 if at least one of a household's coupons is redeemed, and 0 otherwise.
  The researcher will distribute coupons at the household survey. A subject is eligible for a coupon if s/he is not reported HIV+ and has not had an HIV test within 3 months before the visit. A coupon for an adult will be distributed to themselves. A coupon for a child (age <18) will be distributed to their primary guardian. Each coupon has a value of 50Mts (0.83 USD) and is valid for 14 days.
  To redeem a coupon, a coupon holder must show up in the designated clinic and provide proof of testing dated within the coupon-validity window.
  There is a unique barcode on each coupon to allow the researcher to track the use of each coupon. A coupon will be scanned when distributed and redeemed to link to a subject.
  The analysis sample for this outcome of interest is all households that have received at least one coupon from the researcher.
Indicator for school attendance at the child-level | The time when the research team is conducting the school visit, which lasts 4 to 8 hours in each school
  This is an individual-level binary variable. It takes value 1 if a school-aged child (6 -17 years of age) is physically present at school on the date the research staff conducts an unannounced school visit; it takes the value of 0 otherwise.
  The research team will make an unannounced school visit to check the attendance of all school-aged children in the study sample. All school-aged children will be checked regardless of his or her guardian-reported school attendance status. The study team will visit all public primary and secondary schools located in the study community. All unannounced visits will happen on regular school days. Each child will be checked in all neighboring schools. Each child will only be checked once in one school.
  The analysis sample of this outcome of interest is all school-aged children living in the study households.

CONTACTS AND LOCATIONS:
Locations (1):
- Lessitala Consultoria e Servicos, Beira, Sofala, Mozambique